CLINICAL TRIAL: NCT03997708
Title: Mediterranean Diet Adjusted to Low FODMAP Diet (MED-LFD) vs NICE Guidelines for Improving IBS Symptoms: a New Approach for Managing IBS
Brief Title: A Mediterranean Approach to Low FODMAP Diet (MED-LFD) for Managing IBS Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: Department of Gastroenterology, Central Clinical School, Monash University (Unknown)
Responsible Party: Principal Investigator, Arezina Kasti, Head of Dpt of Clinical Nutrition, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ΕΒΔ435/19-06-2018
Record Dates: First submitted 2019-06-14; First posted 2019-06-25 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS; Quality of life; FODMAP; Mediterranean Diet; Clinical Nutrition; low FODMAP
MeSH Terms: interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): MED-LFD Diet (diet A) for 2 - 6 weeks. After this period there will be a reintroduction phase protocol that will last 6 - 8 weeks.
  Interventions: Other: Med-LFD
- Group B (Active Comparator): Diet according to guidelines from the National Institute for Health and Care Excellent (NICE) Managing IBS (diet B) for 4 weeks.
  Interventions: Other: Nutritional Guidelines of the British National Institute for Health and Care Excellence (NICE) Managing IBS

INTERVENTIONS:
Other: Med-LFD — All participants of this group at phase 1 (elimination phase), will initially follow the Med- LFD (2-6 weeks). At phase 2 (reintroduction phase), patients will gradually reintroduce foods rich in FODMAPs (6-8 weeks) and test their tolerance. At phase 3 (maintenance phase), following the reintroduction of foods rich in FODMAPs, patients will follow an individualized diet based on their personal tolerance (a combination of high and low FODMAPs).
  Arms: Group A
Other: Nutritional Guidelines of the British National Institute for Health and Care Excellence (NICE) Managing IBS — All participants of this group will be informed to follow a diet based on the nutritional guidelines of the British National Institute for Health and Care Excellence (NICE) for Managing IBS for 4 weeks.
  Arms: Group B

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common functional bowel disorder characterized by absence of any organic cause. The vast majority of patients associate their symptoms with specific food consumption, creating the need for developing a new therapeutic approach based on altering the dietary habits. The aim of the study focuses in the comparison of the efficacy of two dietary patterns, the adjusted to the Mediterranean Diet Low FODMAP Diet (MED-LFD) and the nutritional guidelines of the British National Institute for Health and Care Excellence (NICE) Managing IBS.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a functional bowel disorder. Patients associate their symptoms with specific foods consumption, creating the need for developing a new therapeutic approach based on altering the dietary intake of these patients. Low FODMAP Diet is often used as a first-line treatment based on observations showing that short-chain carbohydrates are not adequately absorbed in the small intestine and exacerbate the symptoms of IBS. Additionally, the Mediterranean diet is a cultural heritage representative of all the countries surrounded by the Mediterranean Sea, described as a diet rich in herbal foods (cereals, fruits, vegetables, legumes, nuts, olives), with olive oil as the main consumption of fats, high to moderate consumption of fish and seafood, moderate consumption of eggs, poultry, dairy products and alcohol and low consumption of red meat. On the other hand, the nutritional recommendations of British National Institute for Health and Care Excellence (NICE) managing IBS were created on the grounds of systematic reviews and are based on dietary and lifestyle modifications about caffeine, alcohol, fizzy drinks, fiber, resistant starch, fruits, sorbitol, oat and linseed consumption, meal patterns, probiotics and physical activity.

The direct aim of the study is to compare the efficacy of two dietary patterns, the MED-LFD and the nutritional recommendations of NICE managing IBS. Efficacy will be assessed based on the severity of symptoms. Additionally, possible improvements in quality of life and relief of symptoms between the two groups will be evaluated. Finally, the collected fecal samples will be used to assess the effect of each intervention on gut microbiota.

The sample was calculated to 108 participants with prespecified statistical power 80%, level of significance α=0.05 and 10% adjustment for non-compliance in each group to detect an increase in the primary outcome measure (standard deviation of outcome=60). The above hypothesis of the means was based in the meta-analysis of Peter Varju, et al. 2017. Patients will be recruited by the Department of Clinical Nutrition, Attikon University General Hospital, where the nutritional intervention will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the Rome IV criteria for IBS (IBS-D, IBS-M, IBS-U)
* Provision of written informed consent.
* Commitment of availability throughout the study period.
* IBS-SSS > 175

Exclusion Criteria:

* Any concomitant disease requiring specialized nutrition (e.g. renal failure, diabetes, celiac disease, cerebrovascular disease of the central nervous system, major surgical cavity).
* Pregnancy.
* Breastfeeding.
* IBS-C (Bristol Scale type 1 - 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Change of symptoms severity pre and post intervention using a specialized questionnaire. | Baseline, 4 - 8 weeks and 6 months post intervention
  IBS- SSS contains 5 specific questions with instructions on how to score them. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from 0 to a maximum score of 100 using a visual analog scale (VAS) with total scores ranging from 0 to 500, with higher scores indicating more severe symptoms. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS. A decrease of 50 points is associated with a clinically meaningful improvement.

SECONDARY OUTCOMES:
Assessment of IBS related quality of life with a specialized questionnaire pre and post intervention between groups. | Baseline, 4 - 8 weeks and 6 months post intervention
  IBS-QOL - a measure that assesses the degree to which IBS interfered with quality of life over the past 30 days. It is a self-report quality of life measure, which includes domains such as dysphoria, interference with activity, body image, health worry, food avoidance, social relation, sexual and relationship issues. Each of them is rated based on the Likert scale from 1 to 5, the higher the score the lower the quality of life is. The overall score ranges between 34 - 170. A decrease of 10 points or more is a significant improvement.
Assessment of general quality of life pre and post intervention between groups | Baseline, 4 - 8 weeks and 6 months post intervention
  12-Item Short Form Survey (SF-12) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective, covering the eight domains of health outcomes: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional & mental health. The items are weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on the questions that range from 0 to 100, with higher score indicating better health.
Adequate relief of symptoms after the intervention. | Once per week
  Adequate relief (IBS-AR) is a single item questionnaire of pain and discomfort. It poses the question "Over the past week have you had adequate relief of your IBS symptoms?", with a positive or negative answer. Adequate relief is defined as 50% positive answers within the study period, for the purposes of the trial.
Assessment of symptoms burden in general pre and post intervention. | Baseline, 4 - 8 weeks and 6 months post intervention
  The GSRS questionnaire was originally developed for dyspeptic patients but was later validated in patients with IBS. The GSRS is a 15-item questionnaire designed to assess common gastrointestinal symptoms. The questionnaire has five subscales, reflux, diarrhea, constipation, indigestion, and abdominal pain, with subscale scores ranging from 1 (no discomfort) to 7 (severe discomfort). Higher scores represent higher symptom burden.
Assessment of anxiety and depression disorders pre and post intervention. | Baseline, 4 - 8 weeks and 6 months post intervention
  The Hospital Anxiety and Depression Scale (HADS) questionnaire is used for the assessment of anxiety and depression symptoms. It's a 14-item scale with seven items for each subscale, anxiety (HADS-A) and depression (HADS-D). Each item is scored on a response scale with four alternatives, ranging between 0 and 3. The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). A final score of 0-7 on each scale indicates that the patient has no symptoms, a score of 8-10 indicates mild symptoms while a score ≥11 indicates severe symptoms of anxiety and depressive disorders.
Evaluation of the effect of interventions on gut microbiota composition between groups. | Baseline, 2 weeks and 6 months post intervention
  Fecal samples will be collected from each participant and stored at -80°C.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Triantafyllou, Study Director — Attikon Hospital
Locations (1):
- Attikon University General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study, please contact with the research team for more information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study is published.
Access Criteria: Not funded research with similar interest.

REFERENCES:
- [Background] Varju P, Farkas N, Hegyi P, Garami A, Szabo I, Illes A, Solymar M, Vincze A, Balasko M, Par G, Bajor J, Szucs A, Huszar O, Pecsi D, Czimmer J. Low fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) diet improves symptoms in adults suffering from irritable bowel syndrome (IBS) compared to standard IBS diet: A meta-analysis of clinical studies. PLoS One. 2017 Aug 14;12(8):e0182942. doi: 10.1371/journal.pone.0182942. eCollection 2017. PMID 28806407
- [Background] Dalrymple J, Bullock I. Diagnosis and management of irritable bowel syndrome in adults in primary care: summary of NICE guidance. BMJ. 2008 Mar 8;336(7643):556-8. doi: 10.1136/bmj.39484.712616.AD. No abstract available. PMID 18325967
- [Derived] Kasti AN, Katsas K, Pavlidis DE, Stylianakis E, Petsis KI, Lambrinou S, Nikolaki MD, Papanikolaou IS, Hatziagelaki E, Papadimitriou K, Kapolos J, Muir JG, Triantafyllou K. Clinical Trial: A Mediterranean Low-FODMAP Diet Alleviates Symptoms of Non-Constipation IBS-Randomized Controlled Study and Volatomics Analysis. Nutrients. 2025 Apr 30;17(9):1545. doi: 10.3390/nu17091545. PMID 40362860
- [Derived] Kasti AN, Katsas K, Petsis K, Lambrinou S, Synodinou KD, Kapetani A, Smart KL, Nikolaki MD, Halvatsiotis P, Triantafyllou K, Muir JG. Is the Mediterranean Low Fodmap Diet Effective in Managing Irritable Bowel Syndrome Symptoms and Gut Microbiota? An Innovative Research Protocol. Nutrients. 2024 May 23;16(11):1592. doi: 10.3390/nu16111592. PMID 38892525